CLINICAL TRIAL: NCT01254812
Title: Changes on Pulmonary Function After Application of a Bilateral-dual TAP-block
Brief Title: Does the Application of a Bilateral-dual Transverse Abdominal Plane (TAP)Block Have an Influence on Lung Function?
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christian Maschmann, MD, Bispebjerg Hospital
Other Study IDs: H-2-2010-080
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Post Operative Pain
Keywords: pulmonary function; BD-TAP-block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bilateral dual TAP-block
- Placebo Bilateral dual TAP-block

SUMMARY:
TAP-block (Transverse Abdominal Plane) block is a method of regional anesthesia used after abdominal surgery. The method is often applied ultra-sound guided.

In our department, the so-called bilateral dual TAP-block (BD-TAP-block) has been developed. This includes injection of local anesthetics at four sites on the abdominal wall, aiming at the best possible spread of the nerve block.

Clinical experience shows satisfying results on pain relieve using the nerve block, i.e the sensory nerves of the abdominal wall are successfully blocked. However, to our knowledge, clinical investigations regarding the effect on the muscles of the abdominal wall has never been executed.

Patients with chronic lung diseases, who are prone to catch pneumonia post surgery, may have to be able to use accessory muscle groups to prevent pulmonary phlegm stagnation. Therefore it would be inappropriate if the motor nerves supplying these muscles were too, affected by the nerve block.

Our clinical experience has so far not given us suspicion or indication that the motor nerves become blocked, although these nerves are situated in the same muscle layer as the sensory branches.

Hence the investigators would like to examine on healthy, male subjects, whether application of a bilateral-dual TAP-block effects their ability to perform peak-flow and inspiratory and expiratory pressure. Our study hypothesis is:

There is no clinically relevant difference in the spread of results of pulmonary tests (peak flow et.c.) before and after application of bilateral dual TAP-block.

ELIGIBILITY:
Inclusion Criteria:

* No history of asthma
* Young male
* Has to be able to conduct lung function examination and the application of abdominal nerve block

Exclusion Criteria:

* History of asthma

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young (18-45 yrs), healthy males with no history of lung diseases.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | 1 hour after application of the BD-TAP-block

SECONDARY OUTCOMES:
Expiratory/Inspiratory pressure | 1 hour after application of the BD-TAP-block

CONTACTS AND LOCATIONS:
Overall Officials: Christian P. Maschmann, MD, Study Director — Bispebjerg Hospital; Maria Petersen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Dept. of Anesthesiology, Copenhagen NV, Denmark